CLINICAL TRIAL: NCT05460221
Title: Antihypertensive and Cardioprotective Clinical Evaluation of a Functional Olive Oil Enriched in Bioactive Compounds From the Olive Tree
Brief Title: Antihypertensive and Cardioprotective Evaluation of a Functional Olive Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Complejo Hospitalario Universitario de Santiago (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, María Dolores Mesa García, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEDKIDS_HTA; IDI-20190985 (Other Grant/Funding Number: proyectos CIEN (CDTI))
Record Dates: First submitted 2022-03-07; First posted 2022-07-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
Keywords: Extra virgin olive oil; Polyphenols; Triterpenic acids; Hipertensive children
MeSH Terms: conditions — Hypertension | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimized oil group (Active Comparator): Each participant will consume 25 mL/day during 6 months of an Optimized extra virgin olive oil obtained by mixing different varieties of oils rich in bioactive compounds (it contains approx. 490 ppm of bioactive compounds).
  Interventions: Dietary Supplement: Optimized oil group
- Functional oil group (Experimental): Each participant will consume 25 mL/day during 6 months of a Functional olive oil prepared with the same Optimized oil and enriched with triterpenic acids obtained from the olive tree (approx. 490 ppm of polyphenols and 380 ppm of triterpenic acids).
  Interventions: Dietary Supplement: Functional oil group
- Control Group (Placebo Comparator): Each participant will consume 25 mL/day during 6 months of a Control extra virgin olive oil prepared from the same Optimized oil washed to eliminate bioactive compounds (approx. 125 ppm of polyphenols).
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Optimized oil group — This is a controlled parallel study. The patient will receive 25 mL/day of three different types of olive oils with different amouns of bioactive compounds from the olive tree, that must be consumed throughout the day at breakfast or snack (depending on the habits of each child). The doses that they do not take must be returned to the hospital staff to assess adherence to the intervention. The families will receive the same type of oil so that they can cook with it during the study period.
  The control oil will be the same extra virgin olive oil washed to decrease bioactive components (approx. 125 ppm).
  The intervention will take place for 6 months.
  Arms: Optimized oil group
Dietary Supplement: Functional oil group — This is a controlled parallel study. The patient will receive 25 mL/day of three different types of olive oils with different amouns of bioactive compounds from the olive tree, that must be consumed throughout the day at breakfast or snack (depending on the habits of each child). The doses that they do not take must be returned to the hospital staff to assess adherence to the intervention. The families will receive the same type of oil so that they can cook with it during the study period.
  The control oil will be the same extra virgin olive oil washed to decrease bioactive components (approx. 125 ppm).
  The intervention will take place for 6 months.
  Arms: Functional oil group
Dietary Supplement: Control group — This is a controlled parallel study. The patient will receive 25 mL/day of three different types of olive oils with different amouns of bioactive compounds from the olive tree, that must be consumed throughout the day at breakfast or snack (depending on the habits of each child). The doses that they do not take must be returned to the hospital staff to assess adherence to the intervention. The families will receive the same type of oil so that they can cook with it during the study period.
  The control oil will be the same extra virgin olive oil washed to decrease bioactive components (approx. 125 ppm).
  The intervention will take place for 6 months.
  Arms: Control Group

SUMMARY:
The general objective of this study is to evaluate the effect of a nutritional intervention with an extra virgin olive oil (EVOO) rich in bioactive compounds (polyphenols) and a functional oil of adequate organoleptic quality, prepared with the same EVOO rich in polyphenols and also enriched in triterpenic acid compounds from the olive itself, and demonstrate its antihypertensive and cardioprotective effect in children and adolescents (between 6-18 years) at risk of untreated hypertension.

DETAILED DESCRIPTION:
A clinical study of nutritional intervention, randomized, adjusted by randomization blocks that consider age and sex, and parallel duration of 6 months, in 75 subjects (25 per randomization group) is proposed. The study will be carried out at the UGC of Pediatrics of the Reina Sofía University Hospital in Córdoba, as well as at the Institute of Nutrition and Food Technology of the University of Granada.

The effects of an optimized oil rich in polyphenols and obtained by mixing varieties rich in said bioactive compounds (approx. 490 ppm), and a functional oil prepared with the same optimized oil and enriched with triterpenic acids obtained from the olive itself (approx. 490 ppm of polyphenols and 380 ppm of triterpenic acids). The study will be carried out in pediatric patients with high levels of untreated blood pressure, in which the effect of oils on blood pressure and their action on biomarkers of cardiovascular risk and on the intestinal microbiota will be evaluated, depending on the genotype specific to each subject. In addition, the presence of minor olive oil compounds present in the plasma will be analyzed (metabolomic analysis). In this way, at the end of the project, verified scientific information will be available on the enriched product and its effects on cardiovascular protection, and on possible mechanisms of action, as well as on its palatability and acceptance.

The general objective of this study is to evaluate the effect of a nutritional intervention with an EVOO rich in bioactive compounds (polyphenols) and a functional oil of adequate organoleptic quality, prepared with the same EVOO rich in polyphenols and also enriched in triterpenic acid compounds from the olive itself, and demonstrate its antihypertensive and cardioprotective effect in children and adolescents (between 6-18 years) at risk of untreated hypertension.

As specific objectives will be determined:

* To evaluate the effect of olive oils on blood pressure levels
* To evaluate the effect of olive oils on the levels of other components of the metabolic syndrome.
* To evaluate the effect of olive oils on the antioxidant defense system
* To evaluate the effect of olive oils on biomarkers of cardiovascular risk, including markers of inflammation and endothelial damage.
* To evaluate the effect of olive oils on the intestinal microbiota.
* To evaluate the effect of olive oils on metabolomic changes in plasma.
* To analyze the specific genotype of each volunteer and its relationship with the clinical effects found.

ELIGIBILITY:
Inclusion Criteria:

Age between 6 and 18 years Percentile levels compatible with arterial hypertension or very high risk (SBP and/or DBP over P90) Without previous medication for hypertension Acceptance to participate by signing the informed consent

Exclusion Criteria:

Children under 6 years of age Absence of hypertension Children who require or receive some type of medication to control blood pressure, glucose levels or dyslipidemia or any probiotic Not to sign the informed consent.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Changes of systolic blood pressure | 0 month; 3 month; 6 month
  Changes on systolic blood pressure will be measured at the beginning, 3 and 6 months after the intervention. It will be measured in a sitting position and after 5 minutes of rest, using an OMRON HEM 705 CP device, with the cuff adapted to each child, on the left arm. Systolic and diastolic blood pressure will be measured in duplicate, and the mean of both measurements will be recorded, in millimeters of mercury.
Change from Baseline Diastolic Blood Pressure at 6 months | 0 month; 3 month; 6 month
  Changes on systolic and diastolic blood pressure will be measured at the beginning, 3 and 6 months after the intervention. It will be measured in a sitting position and after 5 minutes of rest, using an OMRON HEM 705 CP device, with the cuff adapted to each child, on the left arm. Systolic and diastolic blood pressure will be measured in duplicate, and the mean of both measurements will be recorded, in millimeters of mercury.

SECONDARY OUTCOMES:
Change n weight from baseline to 6 months | 0 month; 3 month; 6 month
  Change from baseline weight (kg) at 6 months. For weight assessment, a Tanita 780PMA model precision scale will be used. It will always be carried out with the patient in underwear, standing on the scale in a standard anatomical position without using any extra point of support that could modify the measurement.
  Patients will be measured with the direct reading Harpenden Stadiometer with a wall-mounted indicator counter, measuring 600-2100 mm, approved by the University of London Institute of Child Health; standing on the height rod, without wearing shoes.
Change on body mass index (BMI) from Baseline to 6 months | 0 month; 3 month; 6 month
  To calculate changes in BMI is necessary to determine weight (kilograms) and height (meters).
  The body mass index (BMI) or Quetelet index (Weight/Height²) will be stratified according to the International reference values of Cole and Bellizi to classify obesity.
Change of body composition from Baseline to 6 months | 0 month; 3 month; 6 month
  Bioimpedance test will be performed to assess changes on body composition, with emphasis on fat mass, using a Tanita 780PMA model precision scale.
Dietary intake and eating habits | 0 month; 3 month; 6 month
  Assessment of changes on dietary intake will be evaluated at the beginning, 3 and 6 months after the intervention with three 24-hour reminders separated by at least one week in accordance with the EFSA recommendations for this type of study, all of them previously validated. At the beginning of the study, a questionnaire on the frequency of food consumption will be carried out.
Physical activity | 0 month; 3 month; 6 month
  Assessment of changes on physical activity will be assessed at the beginning, 3 and 6 months after the intervention through the PAQ-C Physical Activity questionnaire
Sedentary activities | 0 month; 3 month; 6 month
  Assessment of the level of sedentary activities will be evaluated at the beginning, 3 and 6 months after the intervention through an ad hoc questionnaire on time spent watching television and use of computers, video games and consoles, validated for young children and school children, as well as other socioeconomic determinants
Hemogram | 0 month; 3 month; 6 month
  Changes on blood count will be analyzed on an automated analyzer
Blood glucose | 0 month; 3 month; 6 month
  Changes on blood glucose will be analyzed by the glucose oxidase method on an automated analyzer (Roche-Hitachi Modular P and D Autoanalyser; Roche Laboratory Systems, Mannheim, Germany)
Blood insulin | 0 month; 3 month; 6 month
  Changes on plasma insulin will be analyzed by radioimmunoassay (RIA) using an automated microparticle analyzer. (AxSYM; Abbott Laboratories, Abbott Park, IL, USA).
Insulin resistance | 0 month; 3 month; 6 month
  Changes on insulin resistance (IR) will be calculated by homeostatic model assessment of IR (HOMA-IR).
Serum triacylglycerides | 0 month; 3 month; 6 month
  Changes on serum, triglycerides will be measured using an automatic analyzer ( Roche-Hitachi Modular P and D Autoanalyser; Roche Laboratory Systems, Mannheim, Germany).
Serum cholesterol | 0 month; 3 month; 6 month
  Changes on serum total cholesterol, high-density lipoprotein cholesterol (HDLc) and low-density lipoprotein cholesterol (LDLc), as well as Apoprotein A and B, and Lipoprotein A1 will be measured using an automatic analyzer ( Roche-Hitachi Modular P and D Autoanalyser; Roche Laboratory Systems, Mannheim, Germany).
Endothelial function biomarkers in blood | 0 month; 3 month; 6 month
  Simultaneous detection of endothelial adhesion molecules VCAM-1, ICAM, E-selectin and myeloperoxidase will be performed in children's plasma, using MULTIPLEX assay kits and Luminex xMAP detection technology, which allows us to quantitatively determine several biomarkers using a very small amount of sample (25-50 µl of plasma or serum). The HCVD2MAG-67K kit will be used to determine the adhesion molecules.
Antioxidant glutathione reductase activity in red blood cells | 0 month; 3 month; 6 month
  Assessing changes of glutathione reductase activity will be carried out using standardized spectrophotometric methods.
Antioxidant glutathione peroxidase activity in red blood cells | 0 month; 3 month; 6 month
  Assessing changes of glutathione peroxidase activity will be carried out using standardized spectrophotometric methods.
Antioxidant superoxide dismutase activity in red blood cells | 0 month; 3 month; 6 month
  Assessing changes of superoxide dismutase activity will be carried out using standardized spectrophotometric methods.
Antioxidant catalase activity in red blood cells | 0 month; 3 month; 6 month
  Assessing changes of catalase activity will be carried out using standardized spectrophotometric methods.
Antioxidant alpha-tocopherol, beta-carotene, retinol and Coenzyme Q in plasma | 0 month; 3 month; 6 month
  Assessing changes of plasma antioxidants: alpha-tocopherol, beta-carotene, retinol, and coenzyme Q will be analysed by HPLC-MS in one single inyection
Urine endothelin-1 | 0 month; 3 month; 6 month
  Assessing changes of endothelin-1 will be analyzed in plasma using an ELISA kit.
Analysis of oxLDL in plasma | 0 month; 3 month; 6 month
  Assessing changes of oxidized LDL from the baseline to the end of each treatment, by using an ELISA kit
F2-Isoprostanes in urine | 0 month; 3 month; 6 month
  Assessing changes of F2-Isoprostanes will be carried out using an ELISA kit.
8-hydroxy-deoxy-Guanosine in urine | 0 month; 3 month; 6 month
  Assessing changes of 8-hydroxy-deoxy-Guanosine will be carried out using an ELISA kit.
Metagenomics | 0 month; 6 month
  Assessing changes of fecal microbiome profile from the baseline to the end of each treatment. Stool DNA will be isolated with the QIAamp DNA stool mimi kit. Amplification of variable region V3-V1 of 16S gen will be sequenced using the Illunina Next Generation Sequencing MiSeg.
Plasma metabolomic analysis | 0 month; 6 month
  A liquid chromatography platform coupled to a spectrophotometer will be used mass (LC/MS) to determine metabolic profiles by targeted analyses
Urine metabolomic analysis | 0 month; 3 month; 6 month
  A liquid chromatography platform coupled to a spectrophotometer will be used mass (LC/MS) to determine metabolic profiles by targeted analyses
Genotyping | 0 month
  Genotyping of the main candidate genes related to the development of arterial hypertension described in GWAS studies (ACE, ADRB1, AGT, PHACTR1, EDN1, ATP13A3) will be carried out in the Department of Biochemistry and Molecular Biology II of the University of Granada.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA DOLORES MESA GARCIA, Principal Investigator — Universidad de Granada
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofia de Córdoba, Córdoba
  - Universidad de Granada, Granada

IPD SHARING:
Plan to Share IPD: No